CLINICAL TRIAL: NCT03253133
Title: Phase I Study Assessing Safety of Intraperitoneal Chemotherapy in Neoadjuvant Treatment of Peritoneal Carcinomatosis of Colorectal Origin
Brief Title: Assessing Safety of NIPOX in Peritoneal Carcinomatosis of CRC
Acronym: NIPOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC2015/34
Record Dates: First submitted 2016-08-29; First posted 2017-08-17 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin (Experimental): IP neoadjuvant chemotherapy protocol:
  Oxaliplatine will be administered in IP in a total solution of 2L of serum G5%. A continuous infusion pump of Oxycodone would be administered for the entire duration of the intraperitoneal chemotherapy. Perfusion time for the intraperitoneal chemotherapy is estimated but not limited to one and a half hour.
  Intravenous chemotherapy protocol:
  Associated Intravenous (systemic) chemotherapy is administered during IP chemotherapy including at least LVFU2 (5FU-Leucovorin) or FOLFIRI (5FU-Irinotecan) regimens and targeted therapy if needed.
  Interventions: Drug: Oxaliplatin; Drug: LV5FU or Folfiri; Drug: Oxycodone

INTERVENTIONS:
Drug: Oxaliplatin — Dose levels of Oxaliplatin:
  4 dose levels of Oxaliplatin (85, 100, 130 and 160 mg/m²) are planned. 1 dose level is planned (-1 : 70 mg/m²) if DLT is reached at level 1
  Table 1: Dose levels
  Dose Level Dose (mg/m²) Number of patients DL -1 70 mg 3-6 DL 1 * 85 mg 3-6 DL 2 100 mg 3-6 DL 3 130 mg 3-6 DL 4 160 mg 3-6
  * Start level
Drug: LV5FU or Folfiri — Association of chemotherapy by LV5FU or Folfiri according pratician choice
Drug: Oxycodone — Oxycodone

SUMMARY:
This study determine the maximal tolerate dose

DETAILED DESCRIPTION:
This study determine the maximal tolerate dose for the patient treated by intraperitoneal chemotherapy in neoadjuvant treatment of peritoneal carcinomatosis of colorectal origin

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old
2. Histologically confirmed diagnosis of colorectal or appendix cancer
3. Peritoneal carcinomatosis of colorectal origin, presumed unresecable or non-optimally resecable, assessed by imaging (CT scan (Computed Tomography Scanner) and MRI (Magnetic Resonance Imaging)) or during a previous abdominal surgery
4. Peritoneal Carcinomatosis Index > 17
5. Previous adjuvant chemotherapy is allowed
6. One or several lines of chemotherapy are allowed
7. Hemoglobin ≥ 10 g/dL (red blood transfusion is allowed if needed), neutrophils ≥ 1.500/mm3, platelets ≥ 100.000/mm3 and white blood cells > 3000 /mm3
8. Total bilirubin ≤ 1.5 Upper limit of normal (ULN), ALT or AST ≤ 3 ULN
9. Serum creatinine ≤ 1.5 ULN ; Serum calcium ≥ LLN and ≤ 1.2 x UNL ; Serum magnesium ≥ LLN and ≤ 1.2 x UNL ; Kalemia ≥ LLN
10. ECOG (Eastern Cooperative Oncology group) < 1
11. Life expectancy higher than 8 weeks
12. Negative pregnancy test in women of childbearing potential
13. Use of an effective contraceptive method during the whole treatment and up to 6 months after the completion of treatment
14. Patients affiliated to a French Social Security System
15. Signed informed consent (IC) obtained before any study specific procedures

Exclusion Criteria:

1. Serum uracile ≥ 16 ng/ml
2. Extra peritoneal metastatic disease (except ovarian metastases and retroperitoneal nodes)
3. Patients with anesthetic or medical contraindications to surgery
4. Peripheral sensory neuropathy ≥ grade 2 at the time of signing the ICF
5. Patients previously treated with cytoreduction and followed by an intra-peritoneal chemotherapy within the past 6 months.
6. Anticancer therapy (e.g. chemotherapy, radiotherapy, targeted therapy, concomitant systemic immune therapy, or any experimental therapy) within 4 weeks before inclusion
7. History or presence of other cancer within the past 5 years (except adequately treated in situ carcinoma of the cervix and non-melanoma skin cancer)
8. Pregnant or breastfeeding women
9. Known positive test for human immunodeficiency virus (HIV), hepatitis B or C virus or patients with untreated serious infections
10. Participation in another clinical trial within 30 days prior to study entry
11. Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study
12. ECG with a QT/QTc interval higher than 450 ms for men and higher than 470 ms for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | through study completion, an average of 3 year
  To determine:
  - Maximum tolerated dose (MTD),

SECONDARY OUTCOMES:
Area Under the Curve (AUC) | through study completion, an average of 3 year
  To evaluate Long term pharmacokinetic profile of associated targeted agents in tumoral tissue

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Sgarbura, Study Chair — Institut régional du Cancer de Montpellier
Locations (1):
- Institut réginal du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No